CLINICAL TRIAL: NCT04561830
Title: Total Mesorectal Resection With Dissection of the Lateral Pelvic Lymph Nodes in Low Advanced Cancer Rectum Patients; Laparoscopic Versus Open Approach
Brief Title: Open or Laparoscopic Mesolectal Excision in Low Rectum Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, osama khalil, assistant professor, Zagazig University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR 180033-7
Record Dates: First submitted 2020-09-15; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Active Comparator): underwent laparoscopic-assisted excision of mesorectum
  Interventions: Procedure: laparoscopic-assited excision of mesorectum with pelvic lymph nodes excision
- group 2 (Active Comparator): open excision of mesorectum
  Interventions: Procedure: laparoscopic-assited excision of mesorectum with pelvic lymph nodes excision

INTERVENTIONS:
Procedure: laparoscopic-assited excision of mesorectum with pelvic lymph nodes excision — We performed laparoscopic dissection of the lateral pelvic lymph node for thirty patients while we performed open lateral pelvic lymph node dissection for the remaining thirty patients.
  Performed surgical approaches were abdominoperineal resection, internal sphincter resection, and low anterior resection. All performed surgical procedures included lateral pelvic lymphadenectomy in addition to performing total mesorectal excision.
  Choosing whether to perform unilateral or bilateral lymphadenectomy depends on lymph nodes invasion by cancer was on one side or both sides.
  Other Names: open excision of mesorectum with pelvic Lymph nodes excision

SUMMARY:
To compare the open approach and the laparoscopic-assisted approach of dissection of lateral lymph nodes in low advanced rectal cancer patients with clinically suspected nodal metastases in terms of safety, technical feasibility, and patient's oncological outcomes.

DETAILED DESCRIPTION:
the investigators collected data of sixty low advanced cancer rectum patients who underwent either laparoscopic (30 cases) or open total mesorectal excision (30 cases) in addition to lateral pelvic dissection. The duration of operation in the laparoscopically assisted procedure was longer than the open procedure (p=0.003). The postoperative hospital stay time was longer in the open group than in the laparoscopic group (P=0.043). No significant differences between both groups regarding the number of excised lymph nodes, disease recurrence, RFS, or OS rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 20-70 years with
* Sure diagnosis of locally advanced (T3 and T4) adenocarcinoma located in the middle or lower part of the rectum
* Clinical or radiological evidence of lateral pelvic lymph nodes metastases

Exclusion Criteria:

* Patients refused to be included in the study,
* Patients with concurrent primary cancer in other locations
* Patients with recurrent cancer after treatment
* Patients with distant metastasis
* Previously managed for pelvic cancer

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
operative time | during operative time
  time of surgery in minutes
operative complication | durning operative time
  bleed-injury of organs -failed procedure
feasibility of procedure | operative time
  easy or difficult

SECONDARY OUTCOMES:
post operative morbidity | 5 years
  early and late complications
mortality | 5 years
  number of deaths
recurrence | 5 years
  recurrent cases

IPD SHARING:
Plan to Share IPD: No